CLINICAL TRIAL: NCT00388232
Title: Inonu University, The Department of Pulmonary Medicine
Brief Title: Prevalence of COPD: First Epidemiological Data From a Large Region of Turkey
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Other Study IDs: 1-Gunen
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2006-10-16 (Estimated); Status verified 2006-10

CONDITIONS: COPD Prevalance
Keywords: COPD; prevalence; smoke; biomass; occupational; Malatya; Turkey
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The study was designed to obtain some baseline data on COPD in Malatya region of Turkey.

DETAILED DESCRIPTION:
Sixty clusters from urban and rural regions were randomly selected. Ten and seven consecutive houses were included in the study from each urban and rural cluster respectively. A validated questionnaire on epidemiology of COPD was completed for each household over 18 by a pulmonary physician. Each subject performed the standard spirometric measurement and early bronchodilation testing.

ELIGIBILITY:
Inclusion Criteria:

* All households over 18 were included in the study

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1200

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gunen, Associate Professor, Study Chair — Inonu University Department of Pulmonary Medicine